CLINICAL TRIAL: NCT00571012
Title: Aqueous Outflow Facility Changes With Posture
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Deepan Selvadurai MD, Mayo Clinic
Other Study IDs: 07-006662
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: glaucoma; outflow facility; Healthy eye function
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Only one group- A: Healthy young subjects aged 18-45.

SUMMARY:
Intraocular pressure (IOP) varies with body position, with a significant increase occurring from the seated to the supine position. Previous research has indicated that the IOP increase cannot be explained by changes in episcleral venous pressure(blood flow leading away from the eye) alone. As well, previous research has indicated that aqueous flow rate is independent of body position. The purpose of this project was to determine if aqueous humor outflow facility varied with changes in posture.

DETAILED DESCRIPTION:
On the day of the experiment, patients will be asked to maintain a regular schedule and normal activities. This will include avoiding excess caffeine intake, large deviations from normal sleep cycle, or exposure to pharmacologic IOP modifying agents.

Subjects will be seated in standard ophthalmologic examining chairs and reclined into the supine position in a quiet room with subdued lighting for approximately 5 minutes. Anesthesia will be achieved by instilling 3-4 drops of 0.5% proparacaine. The contralateral eye will be patched in an air-tight fashion with an adhesive eye patch to reduce evaporative losses and drying of the cornea. The patient will be asked to keep eyes closed prior to start of measurements. When ready, the patient will be asked to open their eyes and to observe a dim fixation target that will be placed on the ceiling of the room, roughly 6 feet from the patient's eyes. Baseline IOP (Po) will be measured using a pneumatonometer (Model 30 Classic Mentor). Tonography will then be performed using the electronic Schiotz tonometer with a 10g weight in order to obtain a four minute tracing. The procedure will then be repeated on the contralateral eye, with patching of the already tested eye. After this, the patient's chair will the be raised 70 degrees and patient will be asked to hyperextend their neck until their cornea is parallel to the floor. A minimum of 30 minutes will be allowed to elapse, allowing for autonomic, postural and hormonal changes to stabilize. Then a repeat baseline IOP for the sitting position will be taken and another 4 minute tracing will be collected successively in each eye as described above.

Data from the tonometer tracing will be collected electronically and will be exported to a standard Excel file. A smooth curve of best fit will be established through each tonogram once graphed, correcting for oscillations and drift. This curve will help determine the adequacy of the collected sample. Tracings that have a poorly fitted curve might occur for a variety of reasons including patient tenseness and anxiety, uncontrollable tendency to fall asleep and incidental interruptions such as a sudden wave of intestinal peristalsis. Corresponding "Po" values for the initial steady-state IOP and the "C" value for facility of aqueous outflow will be gathered by referring to standard tables and normograms.

The main potential risk of participating in the study is the possibility of corneal abrasion. Previous studies at the Mayo Clinic using the same techniques did not result in any corneal abrasions in over 300 eyes of more than 150 patients. Based on this result, we estimate the risk of a corneal abrasion to be minimal. If a corneal abrasion occurs, the patient will be removed from the study. The patient will be treated with antibiotic drops or ointment and followed until the abrasion has completely healed.

Other minor risks include possible allergic reaction to the anesthetic drops or the adhesive glue. As with any medication, allergic reactions are a possibility. However, these will be the same drops used in routine clinical practice, and allergic reaction is extremely uncommon.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, aged 18-45.
* Subjects will be given a complete dilated eye exam and an updated medical history will be performed

Exclusion Criteria:

* IOP greater than 22mmHg
* Evidence of glaucomatous optic neuropathy
* Poor fixation
* Nystagmus
* Tropias
* Phorias
* Recent infection
* Corneal scarring preventing reliable tonometry
* Evidence of pigment dispersion
* Narrow angles
* History of trauma or surgery
* Systemic use of beta blockers or steroids
* Diabetic eye disease, uveitis, high (>6D) myopia or high(>4D) hyperopia.
* Patients with chronic medical conditions(eg: hypertension) will be allowed to participate as long as their medical condition has been under good control over the preceding 12 months.
* Subjects will also need to have good cervical neck malleability and be able to meet the physical needs of the protocol which call for 4 minutes of neck extension.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young volunteers aged 18-45 will be recruited from Mayo Clinic employees and students, and local area residents.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Looking for change in outflow facility with change in position | 4 minutes per position

CONTACTS AND LOCATIONS:
Overall Officials: Deepan Selvadurai, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] GALIN MA, McIVOR JW, MAGRUDER GB. Influence of position on intraocular pressure. Am J Ophthalmol. 1963 Apr;55:720-3. No abstract available. PMID 13960329